CLINICAL TRIAL: NCT06808126
Title: Evaluation of Ocular Surface Tumors Using Anterior Segment Optical Coherence Tomography (OCT)
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Mohamed Abdelrahman Gebaly, residant doctor, Assiut University
Other Study IDs: Ocular Surface Tumors by OCT
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Ocular Surface Tumors
Keywords: Optical Coherence Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ocular Surface Tumors: patients presented with ocular surface lesion suspected to be neoplastic

SUMMARY:
optical coherence tomography (OCT) can scan a range of ocular tissues and take high-resolution image sections during ophthalmic examination..

and recommended as a rapid, informative and quite reliable method of examination to differentiate benign from malignant ocular surface tumors.

The conjunctiva is an anatomical site with a prominent risk of squamous cell carcinoma development, which is a unique biological behavior. The superficial lesion with significant epithelial cell growth usually displays unique data, contributing to unusual ocular tumors.

Anterior segment optical coherence tomography (AS-OCT), as a noninvasive, high-resolution imaging technique, provides crucial morphological and anatomical information in ocular surface tumors via visualizing the layer structure of the cornea and anterior segment, qualifying tumor morphology, and quantifying thickness and extension. AS-OCT can provide valuable information for helping in clinical diagnoses, differential diagnoses, prognoses, and evaluating responses to treatments as a significant imaging tool in ocular surface tumors.

The correct diagnosis and classification of ocular surface tumors are crucial aspects of their proper management.

the aim of the study • To evaluate the imaging characteristics of ocular surface tumors on high-resolution anterior segment optical coherence tomography (ASOCT).

DETAILED DESCRIPTION:
optical coherence tomography (OCT) can scan a range of ocular tissues and take high-resolution image sections during ophthalmic examination..

and recommended as a rapid, informative and quite reliable method of examination to differentiate benign from malignant ocular surface tumors.

The conjunctiva is an anatomical site with a prominent risk of squamous cell carcinoma development, which is a unique biological behavior. The superficial lesion with significant epithelial cell growth usually displays unique data, contributing to unusual ocular tumors.

Anterior segment optical coherence tomography (AS-OCT), as a noninvasive, high-resolution imaging technique, provides crucial morphological and anatomical information in ocular surface tumors via visualizing the layer structure of the cornea and anterior segment, qualifying tumor morphology, and quantifying thickness and extension. AS-OCT can provide valuable information for helping in clinical diagnoses, differential diagnoses, prognoses, and evaluating responses to treatments as a significant imaging tool in ocular surface tumors.

The correct diagnosis and classification of ocular surface tumors are crucial aspects of their proper management.

the aim of the study • To evaluate the imaging characteristics of ocular surface tumors on high-resolution anterior segment optical coherence tomography (ASOCT).

ELIGIBILITY:
Inclusion Criteria:

* all patients presented with ocular surface lesion suspected to be neoplastic

Exclusion Criteria:

* all patients presented with ocular surface lesion proved by pathology not to be neoplastic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presented with ocular surface lesion suspected to be neoplastic
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
the accuracy of oct | baseline
  the accuracy of oct in diagnosis of Ocular Surface Tumors

IPD SHARING:
Plan to Share IPD: Undecided